CLINICAL TRIAL: NCT05412199
Title: Evaluation of the Acute Effects of Graston, Percussion Massage Therapy, and Dynamic Stretching on Balance, Flexibility, and Performance Parameters in Individuals With Hamstring Tightness.
Brief Title: Which Technique is More Effective for People With Hamstring Tightness in Terms of Balance, Flexibility, and Performance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-2867
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Sports Physical Therapy; Musculoskeletal Diseases or Conditions
Keywords: Hamstring Tightness; Hamstring; IASTM; Graston; Percussion Massage Therapy; Vibration; Dynamic Stretching; Balance; Flexibility; Performance Parameters
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Percussion Massage Therapy Group (Experimental): The group to which percussion massage therapy will be applied to the posterior leg muscles.
  Interventions: Device: Percussion Massage Therapy
- Graston (IASTM) Group (Experimental): The group in which instrument-assisted soft tissue mobilization will be applied to the posterior leg muscles.
  Interventions: Device: Graston
- Dynamic Stretching Group (Experimental): The group to which dynamic stretching exercises will be applied to the posterior leg muscles.
  Interventions: Other: Dynamic Stretching

INTERVENTIONS:
Device: Percussion Massage Therapy — Individuals in the percussion massage therapy group will get 3 minutes of percussion massage therapy on the hamstring and gastrocnemius muscles along the origo-insertion in the mid-frequency range.
  Arms: Percussion Massage Therapy Group
Device: Graston — Instrument-assisted soft tissue mobilization will be used on the hamstring and gastrocnemius muscles along the 5-minute origo insertion line in the Graston group.
  Other Names: IASTM
  Arms: Graston (IASTM) Group
Other: Dynamic Stretching — Dynamic stretching exercises for the hamstring and gastrocnemius muscles will be performed in the dynamic stretching exercise group.
  Arms: Dynamic Stretching Group

SUMMARY:
Percussion massage therapy has gained popularity in the therapeutic and athletic communities over the past few years. Percussion massage therapy devices are extremely convenient to use, both for self-administration and by a physiotherapist. Percussion massage therapy in deep and superficial tissues; is used in many areas such as reducing pain, increasing blood circulation, improving scar tissue, reducing lactate level and muscle spasms, increasing lymphatic flow, inhibiting Golgi reflex, increasing range of motion, and is frequently used today. Vibratory massage techniques have been shown in many studies to improve joint range of motion and muscular strength. It has been argued that there aren't enough studies on this topic in the literature. Specially tailored treatments are utilized in the clinic to reduce injury frequency, improve muscular performance, and increase the flexibility of musculotendinous components. Various stretching methods are used to increase muscle length. Athletes use stretching exercises to improve joint range of motion and long-term performance. Furthermore, it is incorporated in the warm-up period of athletes' training plans to prepare for an activity or to cool down after an applied exercise. Many studies using the dynamic stretching approach have found that dynamic stretching exercises performed before an activity or a sport have a positive effect on performance and flexibility parameters. Instrument-assisted soft tissue mobilization (IASTM) is a treatment method used to reduce pain, improve joint range of motion, and mobilize soft tissue using specially designed stainless steel instruments based on the principles developed by James Cyriax. The removal of scar tissue is one of the most important goals of IASTM. Microvascular bleeding occurs with localized inflammation as a result of IASTM application, nutrient and oxygen flow is delivered, fibroblast migration increases and the healing process begins again. At the same time, secondary collagen synthesis begins and is rearranged, which allows the regeneration of the injured tissue. As a result, it treats scar tissue, adhesions, and adhesions in the fascia. IASTM is a very effective approach in fascia tissue and is widely used to offer a mobilizing stimulus in the treatment of myofascial problems.

DETAILED DESCRIPTION:
However, when the literature is reviewed, studies investigating the acute effects of instrument-assisted soft tissue mobilization, percussion massage therapy, and dynamic stretching exercises on performance parameters and functionality are limited. Based on all this information, it was aimed to investigate the acute effects of percussion massage therapy, stretching exercises, and Graston soft tissue mobilization on jumping, running performance, balance, and functional reaching parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are at a level to be able to perform a performance test
2. With hamstring muscle tightness
3. Those who have not undergone orthopedic surgery from any region
4. Individuals who do not have a professional sports background

Exclusion Criteria:

1. Trauma history
2. Anatomical deformities and skeletal system fractures
3. Diagnosed orthopedic or rheumatological diseases
4. Being included in a physiotherapy program in the last six months
5. Individuals with pain in any part of the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Sit and Reach Test | from pre-interventional time to post-interventional about 1st hour
  The sit and reach test is one of the linear flexibility tests that helps measure the flexibility of the hamstrings and lower back. It was first described by Wells and Dillon in 1952 and is probably the most widely used flexibility test. It has a simple procedure, is easy to administer, requires minimal skill training to perform, and costs the equipment required to perform the test. It is argued that the hamstrings and lower back should have a good level of flexibility, as they play an important role in health-related fitness. In a sitting position on the floor, the soles of the feet are placed on the sit-and-reach bench with the legs fully stretched. Without bending the legs, reach forward with the fingertips on the table and wait 2 seconds at the end point, and the score is recorded in centimeters.
Y Balance Test | from pre-interventional time to post-interventional about 1st hour
  Y Balance Test (YBT) is a functional test that requires strength, flexibility, neuromuscular control, balance, stability, and range of motion (ROM). As an integral part of Functional Movement Systems (FMS), YBT is a thoroughly researched test to test and simultaneously demonstrate an individual's functional symmetry of motor control. YDT gives us the function of each central extremity that is under the weight of a quarter of the body. Six application trials are conducted before the application of this test. The maximum reach analysis in each direction is then performed using three trials in three directions for each leg. Standing on one foot on the midfoot plate with the most distal aspect of the athletic shoe at the baseline, the person being examined stands. The subject is instructed to reach anterior, posteromedial, and posterolateral directions with the free extremity relative to the stance foot while maintaining the single-leg stance, and the distance traveled is measured.

SECONDARY OUTCOMES:
Horizontal Jump Test | from pre-interventional time to post-interventional about 1st hour
  On a flat surface, a starting line is drawn. From the starting line forward, a tape measure is set on the floor, and the athletes are instructed to stand with the tips of both toes pointed towards the back of the previously decided line. The distance jumped is measured in centimeters after the athletes are instructed to bend their knees while keeping their arms parallel to the floor and knees, and to jump as far forward as possible by swinging their arms and legs fast.
Illinois Test | from pre-interventional time to post-interventional about 1st hour
  A test track is set up with three cones lined up in a straight line at intervals of 5 meters(m) in width, 10m in length, and 3.3m in the middle part. The course consists of a 40m straight and a 20m slalom between cones, with 180º bends every 10 meters. Before the test, the subjects are allowed to make 3-4 attempts at low tempo after the introduction of the track and necessary explanations. After that, the subjects are made to do warm-up and stretching exercises for 5-6 minutes at a low tempo that they determine. The test subjects exit the starting line of the test track in a prone position, with their hands at shoulder level in touch with the ground. The time it takes to complete the track is measured in seconds. The test is done two times with full rest between each time, with the better value being recorded.

CONTACTS AND LOCATIONS:
Overall Officials: BURAK MENEK, PhD, Principal Investigator — Medipol University; UMUT İSLAM TAYBOĞA, RA, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)